CLINICAL TRIAL: NCT01785537
Title: Multicentric 5-year Follow-up Study to Assess the Efficacy of E-cigarettes as a Tool for Smoking Cessation and to Compare the Risk of Smoking-related Diseases Among Electronic and Traditional Cigarette Smokers, and Smokers of Both.
Brief Title: The Efficacy and Safety of Electronic Cigarettes: a 5-year Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Collaborators: University of Roma La Sapienza (Other); Catholic University of the Sacred Heart (Other); University of Turin, Italy (Other); University of Catania (Other); Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Principal Investigator, Lamberto Manzoli, Associate Professor of Epidemiology and Public Health, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Other Study IDs: CHLM001
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Cardiovascular Diseases; Chronic Obstructive Pulmonary Diseases; Cancer of the Lung; Cancer of the Bladder; Cancer of the Stomach
Keywords: e-cigarette smoking; cigarette smoking; cardiovascular disease; hospitalization; chronic obstructive pulmonary diseases; observational study; efficacy; safety
MeSH Terms: conditions — Cardiovascular Diseases; Pulmonary Disease, Chronic Obstructive; Lung Neoplasms; Urinary Bladder Neoplasms; Stomach Neoplasms; Cigarette Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- E-cigarettes only: Smokers of e-cigarettes containing nicotine only (non smoking traditional cigarettes and inhaling at least 50 puffs per week since six or more months). This group will be further split in the secondary analyses: never or former smokers of traditional cigarettes
- Traditional cigarettes only: Smokers of traditional cigarettes only (smokers of at least one traditional cigarette per day since six or more months). This group will be further split in the secondary analyses: recent and older smokers.
- Mixed group: Smokers of both electronic and traditional cigarettes (at least one per day since six or more months). This group will be further split in the secondary analyses: mixed smokers who quit and who did not quit traditional cigarette smoking during follow-up

SUMMARY:
The main aim of this multicentric 5-year follow-up study is to evaluate for the first time the long-term efficacy and safety (in terms of smoking-related serious diseases requiring hospitalization) of e-cigarette smoking, comparing its health effects with those of traditional cigarette smoking and mixed electronic and traditional cigarette smoking.

The study will also permit to evaluate, over a 5-year follow-up, the self-reported quality of life, and the reported adverse events according to current and past smoking habit.

Finally, the study will also explore the long-term adherence to e-cigarette smoking and its efficacy of e-cigarettes in reducing and/or quitting traditional cigarette smoking.

ELIGIBILITY:
Inclusion Criteria:

* resident into the Abruzzo and Lazio Region
* aged between 30 and 75 years;
* smoker of e-cigarettes (inhaling at least 50 puffs per week) containing nicotine since six or more months (E-cigarettes only Group);
* smoker of at least one traditional cigarette per day since six or more months (Traditional cigarettes only Group);
* smoker of both electronic and traditional cigarettes (at least one per day) since six or more months (Mixed Group).

Exclusion Criteria:

* illicit drug use,
* breastfeeding or pregnancy,
* major depression or other psychiatric conditions,
* severe allergies,
* active antihypertensive medication,
* angina pectoris,
* past episodes of major cardiovascular diseases (myocardial infarction, stroke/TIA, congestive heart failure, COPD, cancer of the lung, esophagus, larynx, oral cavity, bladder, pancreas, kidney, stomach, cervix, and myeloid leukemia.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult residents in the Abruzzo and Lazio Region of Italy that are smokers of traditional or electronic cigarettes
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2013-10; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Traditional smoking cessation rate | 5 years
  Percentage of subjects that were current (in TC and Mixed groups) or former (in EC group) smokers reporting sustained smoking abstinence from traditional cigarette smoking at 60 months. Smoking abstinence is defined as complete abstinence from tobacco smoking (not even a puff) for the 30 days period prior to the visit. This outcome will be self-reported and checked using CO analyzer after breath.
Change from baseline in the number of traditional cigarette smoked | 6, 12, 24, 36 and 60 months.
  Change in the average self-reported number of traditional cigarette smoked per day.

SECONDARY OUTCOMES:
Rate of subjects with smoking-related hospitalizations | 5 years
  Percentage of subjects who had a hospital admission for one of the followings: cardiovascular diseases, chronic obstructive pulmonary diseases, cancer of the lung, esophagus, larynx, oral cavity, bladder, pancreas, kidney, stomach, cervix, and myeloid leukemia. Repeated admissions of the same subject will be counted once.
Number of smoking-related hospitalizations | 5 years
  Mean number of hospital admissions for one of the followings: cardiovascular diseases, chronic obstructive pulmonary diseases, cancer of the lung, esophagus, larynx, oral cavity, bladder, pancreas, kidney, stomach, cervix, and myeloid leukemia. Each admissions of the same subject will be counted.
Number of hospitalizations for cardiovascular diseases | 5 years
  Mean number of hospital admissions for cardiovascular diseases. Each admissions of the same subject will be counted.
Number of hospitalizations for smoking-related cancers | 5 years
  Mean number of hospital admissions for cancer of the lung, esophagus, larynx, oral cavity, bladder, pancreas, kidney, stomach, cervix, and myeloid leukemia. Each admissions of the same subject will be counted.
Change from baseline in self-reported quality of life | 6, 12, 24 and 36 months
  Change in the average quality of life according to EuroQol EQ-D3.
Time to hospitalization for cardiovascular diseases, COPD and smoking-related cancer. | 5 year
  Time to hospital admission for one of the followings: cardiovascular diseases, chronic obstructive pulmonary diseases, cancer of the lung, esophagus, larynx, oral cavity, bladder, pancreas, kidney, stomach, cervix, and myeloid leukemia. Repeated admissions of the same subject will be counted once and the subject will be censored at the date of the first admission.
Number of Participants with Adverse Events as a Measure of Safety and tolerability | 5 years
  Self-reported side effects as measured by VAS and a structured report form.
Adherence to e-cigarette smoking | 5 years
  Number of months of continued e-cigarette smoking in groups EC and Mixed.
Time to hospitalization for cardiovascular diseases, COPD and smoking-related cancer. | 3 years
  The primary outcome measure is time to hospital admission for one of the followings: cardiovascular diseases, chronic obstructive pulmonary diseases, cancer of the lung, esophagus, larynx, oral cavity, bladder, pancreas, kidney, stomach, cervix, and myeloid leukemia. Repeated admissions of the same subject will be counted once and the subject will be censored at the date of the first admission.
Time to hospitalization for cardiovascular diseases, COPD and smoking-related cancer. | 2 years
  The primary outcome measure is time to hospital admission for one of the followings: cardiovascular diseases, chronic obstructive pulmonary diseases, cancer of the lung, esophagus, larynx, oral cavity, bladder, pancreas, kidney, stomach, cervix, and myeloid leukemia. Repeated admissions of the same subject will be counted once and the subject will be censored at the date of the first admission.
Rate of subjects with smoking-related hospitalizations | 3 years
  Percentage of subjects who had a hospital admission for one of the followings: cardiovascular diseases, chronic obstructive pulmonary diseases, cancer of the lung, esophagus, larynx, oral cavity, bladder, pancreas, kidney, stomach, cervix, and myeloid leukemia. Repeated admissions of the same subject will be counted once.
Rate of subjects with smoking-related hospitalizations | 2 years
  Percentage of subjects who had a hospital admission for one of the followings: cardiovascular diseases, chronic obstructive pulmonary diseases, cancer of the lung, esophagus, larynx, oral cavity, bladder, pancreas, kidney, stomach, cervix, and myeloid leukemia. Repeated admissions of the same subject will be counted once.
Number of smoking-related hospitalizations | 2 years
  Mean number of hospital admissions for one of the followings: cardiovascular diseases, chronic obstructive pulmonary diseases, cancer of the lung, esophagus, larynx, oral cavity, bladder, pancreas, kidney, stomach, cervix, and myeloid leukemia. Each admissions of the same subject will be counted.
Number of smoking-related hospitalizations | 1 year
  Mean number of hospital admissions for one of the followings: cardiovascular diseases, chronic obstructive pulmonary diseases, cancer of the lung, esophagus, larynx, oral cavity, bladder, pancreas, kidney, stomach, cervix, and myeloid leukemia. Each admissions of the same subject will be counted.
Smoking abstinence | 3 years
  Percentage of subjects reporting sustained smoking abstinence from traditional cigarette smoking. Smoking abstinence is defined as complete abstinence from tobacco smoking (not even a puff) for the 30 days period prior to the visit.
Smoking abstinence | 2 years
  Percentage of subjects reporting sustained smoking abstinence from traditional cigarette smoking. Smoking abstinence is defined as complete abstinence from tobacco smoking (not even a puff) for the 30 days period prior to the visit.
Smoking abstinence | 1 year
  Percentage of subjects reporting sustained smoking abstinence from traditional cigarette smoking. Smoking abstinence is defined as complete abstinence from tobacco smoking (not even a puff) for the 30 days period prior to the visit.
Smoking abstinence | 6 months
  Percentage of subjects reporting sustained smoking abstinence from traditional cigarette smoking. Smoking abstinence is defined as complete abstinence from tobacco smoking (not even a puff) for the 30 days period prior to the visit.
Number of Participants with Adverse Events as a Measure of Safety and tolerability | 3 years
  Self-reported side effects as measured by VAS and a structured report form.
Number of Participants with Adverse Events as a Measure of Safety and tolerability | 2 years
  Self-reported side effects as measured by VAS and a structured report form.
Number of Participants with Adverse Events as a Measure of Safety and tolerability | 1 year
  Self-reported side effects as measured by VAS and a structured report form.
Number of Participants with Adverse Events as a Measure of Safety and tolerability | 6 months
  Self-reported side effects as measured by VAS and a structured report form.
Adherence to e-cigarette smoking | 3 years
  Number of months of continued e-cigarette smoking in groups EC and Mixed.
Adherence to e-cigarette smoking | 2 years
  Number of months of continued e-cigarette smoking in groups EC and Mixed.
Adherence to e-cigarette smoking | 1 year
  Number of months of continued e-cigarette smoking in groups EC and Mixed.
Adherence to e-cigarette smoking | 6 months
  Number of months of continued e-cigarette smoking in groups EC and Mixed.
Traditional and electronic smoking (overall smoking) cessation | 1 year
  Percentage of subjects in all groups reporting sustained smoking abstinence from both traditional and electronic cigarette smoking at 12 months. Smoking abstinence is defined as complete abstinence from tobacco or electronic smoking (not even a puff) for the 30 days period prior to the visit.

CONTACTS AND LOCATIONS:
Overall Officials: Lamberto Manzoli, MD, MPH, Principal Investigator — Department of Medicine and Aging Sciences, University of Chieti, Italy
Locations (1):
- Department of Medicine and Aging Sciences, University of Chieti, Chieti, CH, Italy

REFERENCES:
- [Background] Manzoli L, La Vecchia C, Flacco ME, Capasso L, Simonetti V, Boccia S, Di Baldassarre A, Villari P, Mezzetti A, Cicolini G. Multicentric cohort study on the long-term efficacy and safety of electronic cigarettes: study design and methodology. BMC Public Health. 2013 Sep 24;13:883. doi: 10.1186/1471-2458-13-883. PMID 24063569
- [Result] Manzoli L, Flacco ME, Fiore M, La Vecchia C, Marzuillo C, Gualano MR, Liguori G, Cicolini G, Capasso L, D'Amario C, Boccia S, Siliquini R, Ricciardi W, Villari P. Electronic Cigarettes Efficacy and Safety at 12 Months: Cohort Study. PLoS One. 2015 Jun 10;10(6):e0129443. doi: 10.1371/journal.pone.0129443. eCollection 2015. PMID 26061661
- [Result] Manzoli L, Flacco ME, Ferrante M, La Vecchia C, Siliquini R, Ricciardi W, Marzuillo C, Villari P, Fiore M; ISLESE Working Group. Cohort study of electronic cigarette use: effectiveness and safety at 24 months. Tob Control. 2017 May;26(3):284-292. doi: 10.1136/tobaccocontrol-2015-052822. Epub 2016 Jun 6. PMID 27272748